CLINICAL TRIAL: NCT05630001
Title: A Multicenter, Single Arm, Open-label Trial to Evaluate Efficacy and Safety of Oral, Twice Daily Iptacopan in Adult PNH Patients Who Have Hb≥10 g/dL in Response to Anti-C5 Antibody and Switch to Iptacopan
Brief Title: Single Arm, Open Label Trial With Iptacopan Treatment for 24 Weeks, in Patients on Stable Regimen of Anti-C5 Who Switch to Iptacopan.
Acronym: APPULSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023C12303; 2022-502148-10-00 (Other: EU CT)
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Paroxysmal Nocturnal Hemoglobinuria; iptacopan; single arm open-label; Hb≥10 g/dL in response to anti-C5 antibody; switch to iptacopan; PNH; LNP023
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — iptacopan

STUDY DESIGN:
Intervention Model Description: A multicenter, single arm, open-label trial to evaluate efficacy and safety of oral, twice daily iptacopan in adult PNH patients who have Hb≥10 g/dL in response to anti-C5 antibody and switch to iptacopan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LNP023 200mg b.i.d. (Experimental): Iptacopan (LNP023) at a dose of 200 mg b.i.d. orally
  Interventions: Drug: Iptacopan

INTERVENTIONS:
Drug: Iptacopan — Treatment with iptacopan at a dose of 200 mg b.i.d. will start on the first day (Day 1) and continue for 24 weeks.
  Other Names: LNP023

SUMMARY:
The purpose of the study was to find out if iptacopan is effective and safe in adult patients with Paroxysmal Nocturnal Hemoglobinuria (PNH) who switched from their current standard of care treatment (eculizumab or ravulizumab) to study treatment, iptacopan/LNP023.

DETAILED DESCRIPTION:
This was a multicenter, single-arm, open label trial, with iptacopan treatment for 24 weeks in adult PNH patients.

This study was comprised of two periods:

* A Screening period lasting up to 8 weeks.
* A 24-week open-label, iptacopan Treatment period.

After completion of the treatment period, participants who continued to benefit from the iptacopan treatment based on the study doctor's evaluation were able to join the Roll-over extension study (CLNP023C12001B).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male and female participants ≥ 18 years of age, at the time of ICF signatures and with a diagnosis of PNH confirmed by treating physician.
* Stable regimen (dose and intervals) of anti-C5 antibody treatment (either eculizumab or ravulizumab) for at least 6 months prior to screening
* Mean hemoglobin level ≥10 g/dL
* Vaccination against Neisseria meningitidis and S. pneumoniae infection are required prior to the start of iptacopan treatment.
* If not received previously, vaccination against Haemophilus influenzae infections is recommended, if available and according to local regulations.
* Ability to communicate well with the investigator, to understand and comply with the requirements of the study
* Other protocol -defined inclusion criteria may apply at the end.

Exclusion Criteria:

* Participation in any other investigational drug trial or use of other investigational drugs at the time of enrollment
* Patients requiring red blood cell transfusion in the 6 months prior to screening or during screening
* History of stem cell transplantation or any solid organ transplantation
* Active systemic bacterial, viral (incl. COVID-19) or fungal infection within 14 days prior to study drug administration
* Presence of fever ≥ 38.0 °C (100.4 °F) within 7 days prior to study drug administration
* Human immunodeficiency virus (HIV) infection (known history of HIV or test positive for HIV antibody at Screening)
* A history of recurrent invasive infections caused by encapsulated organisms, e.g. meningococcus or pneumococcus
* Unstable medical condition including, but not limited to, myocardial ischemia, active gastrointestinal bleeding, coexisting chronic anemia unrelated to PNH, or unstable thrombotic event not amenable to active treatment as judged by the investigator at Screening.
* History of cancer of any part of the body within the past 5 years,
* Ongoing drug or alcohol abuse that could interfere with patient's participation in the trial.
* Any medical condition deemed likely to interfere with the patient's participation in the study
* Female patients who are pregnant or breastfeeding, or intending to conceive during the course of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (9):
  - City Of Hope National Med Center, Duarte, California
  - USC Norris Cancer Center, Los Angeles, California
  - Lakes Research, Miami Lakes, Florida
  - Mass Gen Hosp Cancer Center, Boston, Massachusetts
  - University Of Minnesota, Minneapolis, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Prisma Health Upstate, Greenville, South Carolina
  - Huntsman Cancer Institute Univ of Utah, Salt Lake City, Utah
- France (3):
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
- Germany (4):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Ulm
- Italy (2):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Bassano del Grappa, VI
- Novartis Investigative Site, Seoul, Seoul, South Korea
- Novartis Investigative Site, Barcelona, Spain
- Novartis Investigative Site, Istanbul, Fatih, Turkey (Türkiye)
- United Kingdom (2):
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 23 centers; 9 in United States, 4 in Germany, 3 in France, 2 in the United Kingdom, 2 in Italy and one each in Spain, Turkey and Republic of Korea enrolled participants.
Pre-assignment Details: The study consisted of a screening period up to 8 weeks.
Period: Overall Study
Arm/Group | LNP023 200mg b.i.d.
Started | 52
Completed | 51
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35
  Asian | 4
  Not Reported | 9
  Unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Hb Levels as Mean of Visits Between Day 126 and Day 168 Compared to Baseline Tested for Non-inferiority
Description: Change in hemoglobin (Hb) levels as mean of visits between Day 126 and Day 168 compared to baseline.
  Baseline is defined as as the mean of three Hb assessments conducted at the central laboratory: two during screening and the third on Day 1.
  The estimation of change from baseline in Hb levels was handled by the hypothetical strategy where participants were assumed as if they did not receive RBC transfusions while on treatment (RBC transfusions were expected to be rare).
  Assuming that participants had stable Hb levels at study entry, the mean change from baseline in Hb level between Day 126 and Day 168 was expected to be unchanged should participants have continued on anti-C5 treatment. Non-inferiority of iptacopan was therefore tested by the null hypothesis (H0) against the alternate hypothesis (H1) comparing the mean change from baseline in Hb level in iptacopan between Day 126 and Day 168 (μ) to -1 g/dL: H0: μ <= -1, H1: μ > -1.
Time Frame: Baseline, Day 126 to Day 168
Population: Full Analysis Set (FAS) comprised all participants with confirmed eligibility to whom study treatment was assigned. The number of participants analyzed corresponds to the number of subjects who had values at baseline and Day 126 and Day 168.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 51
g/dL | 2.01 [1.74 to 2.29]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d; Test type: Non-Inferiority — Non-inferiority and primary objective was considered met if the lower bound of the estimated two-sided 95% confidence interval (CI) is greater than -1 g/dL; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: Change in Hb Levels as Mean of Visits Between Day 126 and Day 168 Compared to Baseline Tested for Superiority
Description: Change in hemoglobin (Hb) levels as mean of visits between Day 126 and Day 168 compared to baseline.
  Baseline is defined as as the mean of three Hb assessments conducted at the central laboratory: two during screening and the third on Day 1.
Time Frame: Baseline, Day 126 to Day 168
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 51
g/dL | 2.01 [1.74 to 2.29]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d; Test type: Superiority — Superiority and the key secondary objective was considered met if the lower bound of the estimated two-sided 95% CI was > 0 g/dL; p < 0.0001, Mixed Models Analysis

3. Secondary Outcome: Proportion of Hematological Responders to Iptacopan Treatment
Description: Response defined as Hb ≥12 g/dL assessed between visits Day 126 and Day 168 in the absence of RBC transfusions, on three out of four measurements taken at the visits occurring in last six weeks
Time Frame: Day 126 to Day 168
Population: Full Analysis Set (FAS) comprised all participants with confirmed eligibility to whom study treatment was assigned. The number of participants analyzed corresponds to the number of subjects who had values at Day 126 and Day 168.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 51
Proportion of participants | 92.7 [84.6 to 98.1]

4. Secondary Outcome: Proportion of Participants Who Remain Free From Transfusions
Description: Number of participants with absence of administration of packed RBC transfusions between Day 1 and Day 168
Time Frame: Day 1 to Day 168
Population: Full Analysis Set (FAS) comprised all participants with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 52
Proportion of participants | 100.0 [93.1 to 100.0]

5. Secondary Outcome: Change From Baseline in Absolute Reticulocytes Count (ARC) Levels
Description: Change from baseline in ARC levels as mean of visits between Day 126 and Day 168
Time Frame: Baseline, Day 126 to Day 168
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 51
10^9 cells/L | -89.19 [-95.47 to -82.92]

6. Secondary Outcome: Percentage Change From Baseline in Lactate Dehydrogenase (LDH) Levels
Description: Percentage change from baseline in LDH levels as mean of visits between Day 126 and Day 168
Time Frame: Baseline, Day 126 to Day 168
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percent change from baseline in LDH
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 51
Percent change from baseline in LDH | -1.30 [-6.56 to 4.26]

7. Secondary Outcome: Change From Baseline in Treatment Satisfaction Score Using TSQM-9 Questionnaire
Description: Difference in scores of the Treatment Satisfaction Questionnaire for Medication(TSQM-9) between baseline and Day 84 and Day 168 assessed after switching from SoC (anti-C5) to iptacopan.
  TSQM-9 is a patient reported outcomes measure that was designed to assess patients' satisfaction with medication across three domains of effectiveness, convenience and global satisfaction. The TSQM-9 contains 3 questions in each domain. Domain scores range from 0 - 100 with higher scores representing better outcomes for the domain.
Time Frame: Baseline, Day 84 and Day 168
Population: Full Analysis Set (FAS) comprised all participants with confirmed eligibility to whom study treatment was assigned. The number of participants analyzed corresponds to the number of subjects who had values at baseline, Day 84 and Day 168.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 50
score on a scale
  TSQMS1-Effectiveness Day 84 | 15.08 [9.60 to 20.57]
  TSQMS1-Effectiveness Day 168: number analyzed (Participants) | 48
  TSQMS1-Effectiveness Day 168 | 12.54 [5.58 to 19.49]
  TSQMS1-Convenience Day 84 | 20.34 [13.68 to 26.99]
  TSQMS1-Convenience 168: number analyzed (Participants) | 48
  TSQMS1-Convenience 168 | 23.86 [17.62 to 30.10]
  TSQMS1-Global Satisfaction Day 84 | 14.26 [9.79 to 18.72]
  TSQMS1-Global Satisfaction Day 168: number analyzed (Participants) | 48
  TSQMS1-Global Satisfaction Day 168 | 18.53 [12.87 to 24.19]

8. Secondary Outcome: Change From Baseline in Fatigue Score Using FACIT-F Questionnaire
Description: Change from baseline in patient-reported scores for the functional assessment of chronic illness therapy - Fatigue (FACIT-F) collected at Day 84 and Day 168.
  The FACIT-F is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. All FACIT scales are scored so that a high score is better. As each of the 13 items of the FACIT-F scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best.
Time Frame: Baseline, Day 84 and Day 168
Population: Full Analysis Set (FAS) comprised all participants with confirmed eligibility to whom study treatment was assigned. The number of participants analyzed corresponds to the number of subjects who had values at Day 84 and Day 168.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 50
score on a scale
  Day 84 | 4.88 [3.23 to 6.53]
  Day 168: number analyzed (Participants) | 47
  Day 168 | 4.29 [1.74 to 6.85]

9. Secondary Outcome: Percentage of Patients Who Had Breakthrough Hemolysis (BTH) Event
Description: Wilson method is used to calculate the confidence interval for the proportion of patients who had events.
  The breakthrough is defined clinical if either there is a decrease in hemoglobin levels equal to or more than 2 g/dL (compared to the latest assessment) or if patients present signs or symptoms of gross hemoglobinuria, painful crisis, dysphagia or any other significant clinical PNH-related signs & symptoms, in presence of laboratory evidence of intravascular hemolysis.
Time Frame: Up to 168 Days
Population: Full Analysis Set (FAS) comprised all participants with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: Percentage of patients with BTH events
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 52
Percentage of patients with BTH events | 0.00 [0.00 to 0.14]

10. Secondary Outcome: Percentage of Patients Who Had Major Adverse Vascular Events (MAVEs)
Description: A MAVE is defined as: acute peripheral vascular occlusion, amputation (non-traumatic; nondiabetic), cerebral arterial occlusion/cerebrovascular accident, cerebral venous occlusion, dermal thrombosis, gangrene (non-traumatic; nondiabetic), hepatic/portal vein thrombosis (Budd-Chiari syndrome), mesenteric/visceral arterial thrombosis or infarction, mesenteric/visceral vein thrombosis or infarction, myocardial infarction, pulmonary embolus, renal arterial thrombosis, renal vein thrombosis, thrombophlebitis / deep vein thrombosis, transient ischemic attack, unstable angina or other.
Time Frame: Up to 168 Days
Population: Full Analysis Set (FAS) comprised all participants with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: Percentage of patients with MAVEs
Arm/Group | LNP023 200mg b.i.d.
Number analyzed (Participants) | 52
Percentage of patients with MAVEs | 0.00 [0.00 to 0.14]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 7 days post treatment for non-serious AEs and 30 days post treatment for serious AEs if patient did not roll over to REP study, up to a maximum duration of 198 days
Arm/Group | LNP023 200mg b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 2/52
Other Adverse Events (participants affected / at risk) | 25/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 200mg b.i.d. (N=52)
Pyrexia (General disorders and administration site conditions) | 1
Pneumonia bacterial (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 200mg b.i.d. (N=52)
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Fatigue (General disorders and administration site conditions) | 4
Nasopharyngitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 3
Headache (Nervous system disorders) | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT05630001/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT05630001/SAP_001.pdf